CLINICAL TRIAL: NCT06874582
Title: EVALUATION of QUALITY of LIFE, PSYCHOSOCIAL ADAPTATION, and FUNCTIONALITY in SILICONE PROSTHESIS USERS
Brief Title: Evaluation of Individuals with Partial or Finger Amputation After Silicone Prosthesis Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, ESRA ATILGAN, Assoc.Prof.Dr., Medipol University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-10840098-772.02-5247
Record Dates: First submitted 2025-02-25; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Amputation; Quality of Life; Psychosocial Adaptation; Silicone Prosthesis; Functionality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- silicone hand or finger prosthesis users (Active Comparator): The first arm of our study consisted of participants with partial or finger amputation and silicone hand-finger prosthesis.
  Interventions: Device: silicone hand or finger prosthesis
- silicone foot or toe prostheses users (Active Comparator): The second arm of our study consisted of participants with partial or finger amputation and silicone foot-foot toe prosthesis.
  Interventions: Device: silicone foot and foot toe prosthesis

INTERVENTIONS:
Device: silicone hand or finger prosthesis — To the best of the author's knowledge, no previous studies have evaluated and compared customised finger and partial silicone prostheses in both extremities. This feature distinguishes the present study from other studies.
  Arms: silicone hand or finger prosthesis users
Device: silicone foot and foot toe prosthesis — To the best of the author's knowledge, no previous studies have evaluated and compared customised finger and partial silicone prostheses in both extremities. This feature distinguishes the present study from other studies.
  Arms: silicone foot or toe prostheses users

SUMMARY:
Objective: This study aimed to evaluate the psychosocial adaptation, functional capacity, and quality of life of individuals who underwent partial hand or foot amputations after using silicone hand and foot prostheses.

Materials and Methods: The study included 32 patients. Demographic and clinical characteristics of the participants were recorded. Participants were divided into two groups as silicone hand or foot prosthesis users. The Visual Analog Scale (VAS) was used to assess pain levels before and after prosthesis use, the Trinity Amputation and Prosthesis Experience Scales (TAPES) were applied to evaluate functional capacity, and the Nottingham Health Profile (NHP) was used to assess quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Hand and foot amputation.
* Aged between 18 and 60 years
* Active employee
* Able to walk, co-operate, move actively with hands
* Who have been using prosthesis for at least 1 year and have good stump-socket compatibility,
* Literate individuals were determined on a voluntary basis.

Exclusion Criteria:

* Multiple amputations
* Severe neurological or traumatic findings
* Individuals with severe deformity or posture disorder that may lead to loss of gait, balance or function.
* With limitation of movement in the upper extremities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Nottingham Health Profile (NHP) | through study completion, an average of 1 year
  The NHP questionnaire consists of two sections with "Yes-No" responses. The first section includes dimensions such as energy levels, pain, emotional reactions, sleep, social isolation, and physical abilities, while the second section addresses the impact of poor health on daily life, covering areas such as employment, household activities, social life, relationships, sexual life, hobbies, and vacations. The first section's total score ranges from 0-600, with higher scores indicating lower activity. The second section ranges from 0-7, with higher scores indicating lower activity.
Trinity Amputation and Prosthesis Experience Scales (TAPES) | through study completion, an average of 1 year
  The TAPES questionnaire evaluates psychosocial adaptation, functionality, and prosthesis satisfaction. It comprises two main sections with nine subscales. The psychosocial subscales include general adaptation, social adaptation, and restriction adaptation, with each rated on a five-point scale (1: Strongly Disagree to 5: Strongly Agree). Scores range from 5 to 25, with higher scores indicating better adaptation.
Visual Analog Scale(VAS) | through study completion, an average of 1 year
  The VAS was used to measure pain in the stump before and after silicone prosthesis use. They were asked to draw their pain level on a 10 cm scale between 0-10 points as 0=no pain, 10 unbearable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided